CLINICAL TRIAL: NCT00672620
Title: A Randomized, Double-Blind, Parallel-Group, Placebo-Controlled, Active-Referenced, Fixed-Dose Study Comparing the Efficacy and Safety of 2 Doses of Lu AA21004 in Acute Treatment of Adults With Major Depressive Disorder
Brief Title: Efficacy and Safety of Vortioxetine (Lu AA21004) in the Treatment of Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LuAA21004_304; U1111-1114-3497 (Registry Identifier: WHO)
Record Dates: First submitted 2008-05-02; First posted 2008-05-06 (Estimated); Results first posted 2013-12-18 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-10

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Depression; Drug Therapy; Major Depressive Episode
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Vortioxetine; Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Vortioxetine 2.5 mg (Experimental): Vortioxetine 2.5 mg, encapsulated tablets, orally, once daily for up to 8 weeks, then placebo-matching capsules, orally, once daily, for 1 week following the treatment period.
  Interventions: Drug: Vortioxetine
- Vortioxetine 5 mg (Experimental): Vortioxetine 5 mg, encapsulated tablets, orally, once daily for up to 8 weeks, then placebo-matching capsules, orally, once daily, for 1 week following the treatment period.
  Interventions: Drug: Vortioxetine
- Duloxetine 60 mg (Active Comparator): Duloxetine 60 mg, capsules, orally, once daily for up to 8 weeks, then duloxetine 30 mg capsules, orally, once daily for 1 week after the treatment period.
  Interventions: Drug: Duloxetine
- Placebo (Placebo Comparator): Placebo-matching capsules, orally, once daily for up to 9 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vortioxetine — Encapsulated vortioxetine immediate-release tablets
  Other Names: Lu AA21004; Brintellix®
  Arms: Vortioxetine 2.5 mg; Vortioxetine 5 mg
Drug: Duloxetine — Duloxetine capsules
  Other Names: Cymbalta®
  Arms: Duloxetine 60 mg
Drug: Placebo — Placebo-matching capsules
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy and safety of vortioxetine, once daily (QD), in adults with major depressive disorder.

DETAILED DESCRIPTION:
The drug that was tested in this study is called Vortioxetine. Vortioxetine is being tested to treat depression in adults who have major depressive disorder (MDD). This study looked at MDD relief in people who took varying dosages of vortioxetine.

The study enrolled 611 patients. Participants were randomly assigned (by chance, like flipping a coin) to one of the four treatment groups-which remained undisclosed to the patient and study doctor during the study (unless there was an urgent medical need):

* Vortioxetine 2.5 mg
* Vortioxetine 5 mg
* Duloxetine 10 mg
* Placebo (dummy inactive capsule) - this was a capsule that looked like the study drug but had no active ingredient.

All participants were asked to take one capsule at the same time each day throughout the study.

This multi-center trial was conducted in the United States. The overall time to participate in this study was up to 12 weeks. Participants made 8 visits to the clinic, and were contacted by telephone 4 weeks after the last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* Suffers from a major depressive episode as the primary diagnosis according to Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM-IV-TR) criteria.
* The reported duration of the current major depressive episode is at least 3 months.

Exclusion Criteria:

* Has 1 or more the following:

  * Any current psychiatric disorder other than major depressive disorder as defined in the DSM-IV-TR.
  * Current or past history of: manic or hypomanic episode, schizophrenia, or any other psychotic disorder, including major depression with psychotic features, mental retardation, organic mental disorders, or mental disorders due to a general medical condition as defined in the DSM-IV-TR.
  * Any substance disorder (except nicotine and caffeine) within the previous 6 months as defined in the DSM-IV-TR.
  * Presence or history of a clinically significant neurological disorder (including epilepsy).
  * Neurodegenerative disorder (Alzheimer disease, Parkinson disease, multiple sclerosis, Huntington disease, etc).
  * Any Axis II disorder that might compromise the study.
* Has a significant risk of suicide according to the investigator's opinion or has a score ≥5 on item 10 (suicidal thoughts) of the Montgomery Åsberg Depression Rating Scale (MADRS) or has made a suicide attempt in the previous 6 months.
* The current depressive symptoms of the patient are considered by the investigator to have been resistant to 2 adequate antidepressant treatments of at least 6 weeks duration each.
* Has received electroconvulsive therapy within 6 months prior to Screening.
* Is currently receiving formal cognitive or behavioral therapy, systematic psychotherapy, or plans to initiate such therapy during the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 611 (Actual)
Dates: Start 2008-04; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Clinical Science, Study Director — Takeda
Locations (38):
- United States (38):
  - Beverly Hills, California
  - Irvine, California
  - Santa Ana, California
  - Torrance, California
  - Upland, California
  - Bradenton, Florida
  - Coral Springs, Florida
  - Fort Walton Beach, Florida
  - Gainesville, Florida
  - Jacksonville, Florida
  - Maitland, Florida
  - Orlando, Florida
  - South Miami, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Smyrna, Georgia
  - Chicago, Illinois
  - Libertyville, Illinois
  - Oak Brook, Illinois
  - Prairie Village, Kansas
  - Owensboro, Kentucky
  - Baltimore, Maryland
  - Pittsfield, Massachusetts
  - Worcester, Massachusetts
  - Flowood, Mississippi
  - New York, New York
  - Olean, New York
  - Beachwood, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Allenport, Pennsylvania
  - Lancaster, Pennsylvania
  - Memphis, Tennessee
  - Austin, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Seattle, Washington
  - Milwaukee, Wisconsin

REFERENCES:
- [Result] Mahableshwarkar AR, Jacobsen PL, Chen Y. A randomized, double-blind trial of 2.5 mg and 5 mg vortioxetine (Lu AA21004) versus placebo for 8 weeks in adults with major depressive disorder. Curr Med Res Opin. 2013 Mar;29(3):217-26. doi: 10.1185/03007995.2012.761600. Epub 2013 Jan 17. PMID 23252878

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 47 investigative sites in the United States from 10 April 2008 to 30 December 2008.
Pre-assignment Details: Participants with a diagnosis of major depressive disorder were enrolled equally in 1 of 4 treatment groups, once a day placebo, 2.5 mg, 5 mg vortioxetine, or 60 mg duloxetine.
Groups:
- Duloxetine 60 mg: Duloxetine 60 mg, capsules, orally, once daily for up to 8 weeks, then duloxetine 30 mg capsule, orally, once daily for 1 week after the treatment period
Period: Overall Study
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Duloxetine 60 mg
Started | 153 | 153 | 153 | 152
Treated | 151 | 149 | 153 | 150
Completed | 120 | 99 | 122 | 110
Not Completed | 33 | 54 | 31 | 42
Not completed — Adverse Event | 7 | 7 | 12 | 17
Not completed — Lack of Efficacy | 1 | 2 | 2 | 0
Not completed — Noncompliance with Study Drug | 3 | 4 | 0 | 2
Not completed — Protocol Deviations | 5 | 7 | 2 | 5
Not completed — Withdrawal of Consent | 6 | 12 | 5 | 6
Not completed — Lost to Follow-up | 8 | 19 | 8 | 11
Not completed — Reason not Specified | 3 | 3 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Duloxetine 60 mg | Total
Number analyzed (Participants) | 153 | 153 | 153 | 152 | 611
Age Continuous [Mean (Standard Deviation); unit: years] | 42.6 (13.76) | 42.6 (12.85) | 43.1 (13.89) | 42.7 (14.38) | 42.7 (13.70)
Age, Customized [Number; unit: participants]
  ≤55 years | 122 | 127 | 125 | 123 | 497
  >55 years | 31 | 26 | 28 | 29 | 114
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 98 | 106 | 91 | 388
  Male | 60 | 55 | 47 | 61 | 223
Race/Ethnicity, Customized [Number; unit: participants] — Number of participants for whom Race data were available were 153, 153, 151 and 151 respectively.
  participants
    Caucasian (White, including Hispanic) | 121 | 112 | 108 | 111 | 452
    Black | 28 | 35 | 40 | 36 | 139
    Asian | 3 | 3 | 3 | 3 | 12
    American Indian or Alaska Native | 1 | 2 | 0 | 0 | 3
    Native Hawaiian/ Other Pacific Islander | 0 | 1 | 0 | 1 | 2
Race/Ethnicity, Customized [Number; unit: participants] — Number of participants for whom Ethnicity data were available were 153, 153, 152 and 151 respectively.
  participants
    Hispanic/Latino | 35 | 21 | 19 | 28 | 103
    Non-Hispanic/Non-Latino | 118 | 132 | 133 | 123 | 506
Region of Enrollment [Number; unit: participants]
  United States | 153 | 153 | 153 | 152 | 611
Weight [Mean (Standard Deviation); unit: kg] | 84.22 (20.144) | 85.08 (24.126) | 88.61 (25.779) | 87.44 (20.695) | 86.34 (22.823)
Height [Mean (Standard Deviation); unit: cm] | 168.98 (9.141) | 169.50 (9.385) | 167.98 (9.833) | 170.37 (9.624) | 169.21 (9.515)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.58 (7.263) | 29.48 (7.479) | 31.38 (8.846) | 30.14 (6.773) | 30.15 (7.649)
Smoking Classification [Number; unit: participants]
  Never smoked | 72 | 81 | 87 | 75 | 315
  Current smoker | 47 | 42 | 45 | 36 | 170
  Ex-smoker | 34 | 30 | 21 | 41 | 126
Alcohol consumption [Number; unit: participants]
  Never | 50 | 49 | 48 | 49 | 196
  Once monthly or less often | 56 | 49 | 62 | 51 | 218
  Once per week | 23 | 26 | 23 | 21 | 93
  2-to-6 times/week | 22 | 20 | 17 | 28 | 87
  Daily | 2 | 9 | 3 | 3 | 17
24-item Hamilton Depression Scale total score [Mean (Standard Deviation); unit: scores on a scale] — The 24-item Hamilton Depression Scale (HAM-D24) is a clinician-rated 24-item scale for assessing the severity of depression symptoms. The scores for each item range from 0 to 4 or 0 to 2, where 0 represents no symptoms. The rating is based on the past 7 days prior to the time of assessment. The total score ranges from 0 to 74, where a higher score indicates a greater depressive state.
  scores on a scale | 29.5 (6.05) | 29.8 (5.42) | 29.8 (5.58) | 28.7 (5.08) | 29.5 (5.55)
Montgomery Åsberg Depression Rating Scale (MADRS) total score [Mean (Standard Deviation); unit: scores on a scale] — The Montgomery Åsberg Depression Rating Scale (MADRS) is a depression rating scale consisting of 10 items, each rated 0 to 6. The 10 items represent the core symptoms of depressive illness. The overall score ranges from 0 (symptoms absent) to 60 (severe depression).
  scores on a scale | 30.0 (4.39) | 29.8 (4.61) | 30.1 (4.51) | 29.4 (4.31) | 29.8 (4.45)
Hamilton Anxiety Scale Total Score [Mean (Standard Deviation); unit: scores on a scale] — Hamilton Anxiety Scale (HAM-A) is an anxiety rating scale consisting of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behavior at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total scores range from 0 to 56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe. Total scores above 30 are rare, but indicate very severe anxiety.
  scores on a scale | 18.8 (5.53) | 19.3 (5.22) | 18.7 (5.74) | 17.4 (5.47) | 18.5 (5.53)
Clinical Global Impression - Severity scale score [Mean (Standard Deviation); unit: scores on a scale] — The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale where the clinician rates the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis on the following scale: 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill.
  scores on a scale | 4.5 (0.62) | 4.6 (0.62) | 4.6 (0.65) | 4.5 (0.67) | 4.5 (0.64)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the 24-item Hamilton Depression Scale Total Score at Week 8
Description: The HAM-D24 is a clinician-rated 24-item scale for assessing the severity of depression symptoms. The scores for each item range from 0 to 4 or 0 to 2, where 0 represents no symptoms. The rating is based on the past 7 days prior to the time of assessment. The total score ranges from 0 to 74 where a higher score indicates a greater depressive state. Least squares (LS) means were from an Analysis of Covariance (ANCOVA) model with terms for treatment and center as factors and the Baseline rank value as a covariate.
Time Frame: Baseline and Week 8
Population: The full analysis set (FAS) included all randomized patients who received at least 1 dose of study drug and had at least 1 valid postbaseline value for assessment of primary efficacy. Last observation carried forward (LOCF) was used.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Duloxetine 60 mg
Number analyzed (Participants) | 149 | 146 | 153 | 149
scores on a scale | -10.50 (0.757) | -12.04 (0.744) | -11.08 (0.737) | -13.47 (0.750)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 5 mg; All statistical tests were 2-sided with 95% confidence intervals (CIs), and with P-values evaluated at the 5% significance level (ie, statistical significance if P<0.05). To control for multiplicity, a pre-specified sequential testing procedure was applied to compare 5 mg and 2.5 mg vortioxetine to placebo; as soon as an endpoint was non-significant at 0.05, the testing procedure stopped for all subsequent endpoints; Test type: Superiority or Other; p = 0.577, ANCOVA — Pre-specified sequential statistical testing procedure indicates that when p-value >0.05, hierarchical testing stops and for subsequent endpoints in the sequence a nominal p-value is provided; ANCOVA with treatment and center as fixed factors, baseline HAM-D24 as covariate; LS Mean Difference = -0.58, 95% CI 2-sided [-2.61 to 1.46], Standard Error of Mean 1.036
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 2.5 mg; Test type: Superiority or Other; p = 0.138, ANCOVA; ANCOVA with treatment and center as fixed factors, baseline HAM-D24 as covariate; LS Mean Difference = -1.54, 95% CI 2-sided [-3.58 to 0.50], Standard Error of Mean 1.038
Statistical Analysis 3: Comparison: Placebo vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.005, ANCOVA; ANCOVA with treatment and center as fixed factors, baseline HAM-D24 as covariate; LS Mean Difference = -2.96, 95% CI 2-sided [-5.02 to -0.91], Standard Error of Mean 1.047

2. Secondary Outcome: Change From Baseline in the 24-item Hamilton Depression Scale Total Score at Other Weeks Assessed
Description: The HAM-D24 is a clinician-rated 24-item scale for assessing the severity of depression symptoms. The scores for each item range from 0 to 4 or 0 to 2, where 0 represents no symptoms. The rating is based on the past 7 days prior to the time of assessment. The total score ranges from 0 to 74 where a higher score indicates a greater depressive state. LS means were from an ANCOVA model with terms for treatment and center as factors and the Baseline rank value as a covariate.
Time Frame: Baseline and Weeks 1, 2, 4, and 6
Population: Full analysis set; LOCF was used. "n" indicates the number of patients included in the analysis at each time point.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Duloxetine 60 mg
Number analyzed (Participants) | 149 | 146 | 153 | 149
scores on a scale
  Week 1 (n=142, 143, 150, 147) | -5.12 (0.515) | -5.44 (0.497) | -5.28 (0.491) | -5.66 (0.500)
  Week 2 (n=149, 146, 153, 149) | -7.19 (0.567) | -7.95 (0.557) | -7.99 (0.552) | -8.42 (0.562)
  Week 4 (n=149, 146, 153, 149) | -9.39 (0.663) | -9.94 (0.651) | -8.96 (0.645) | -10.88 (0.657)
  Week 6 (n=149, 146, 153, 149) | -10.43 (0.706) | -11.21 (0.694) | -10.97 (0.687) | -12.78 (0.700)

3. Secondary Outcome: Percentage of Responders in HAM-D 24 Total Score by Study Visit
Description: A responder is defined as a participant with a ≥50% decrease from Baseline in HAM-D24 total score. The HAM-D24 is a clinician-rated 24-item scale for assessing the severity of depression symptoms. The scores for each item range from 0 to 4 or 0 to 2, where 0 represents no symptoms. The rating is based on the past 7 days prior to the time of assessment. The total score ranges from 0 to 74, where a higher score indicates a greater depressive state.
Time Frame: Baseline and Weeks 1, 2, 4, 6 and 8.
Population: Full analysis set; LOCF was used. "n" indicates the number of patients included in the analysis at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Duloxetine 60 mg
Number analyzed (Participants) | 149 | 146 | 153 | 149
percentage of participants
  Week 1 (n=142, 143, 150, 147) | 9.2 | 8.4 | 8.7 | 10.2
  Week 2 (n=149, 146, 153, 149) | 15.4 | 17.1 | 17.6 | 22.1
  Week 4 (n=149, 146, 153, 149) | 26.2 | 30.8 | 24.2 | 34.9
  Week 6 (n=149, 146, 153, 149) | 32.9 | 37.7 | 37.3 | 47.0
  Week 8 (n=149, 146, 153, 149) | 32.2 | 41.1 | 37.9 | 51.0

4. Secondary Outcome: Percentage of Participants With a Sustained Response in HAM-D24
Description: A sustained response is defined as a ≥ 20% decrease from Baseline in HAM-D24 total score obtained at Week 1 and sustained through Week 7 and at least 50% decrease from Baseline at Week 8.
Time Frame: Baseline to Week 8
Population: Full analysis set with available data.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Duloxetine 60 mg
Number analyzed (Participants) | 149 | 146 | 153 | 149
percentage of participants | 12.1 | 15.8 | 17.0 | 21.5

5. Secondary Outcome: Percentage of Participants in MADRS Remission at Week 8
Description: Remission is defined as a participant with a Montgomery Åsberg Depression Rating Scale (MADRS) total score ≤10. The MADRS is a depression rating scale consisting of 10 items, each rated 0 to 6. The 10 items represent the core symptoms of depressive illness. The overall score ranges from 0 (symptoms absent) to 60 (severe depression). Decrease in the total score or on individual items indicates improvement.
Time Frame: Week 8
Population: Full analysis set; LOCF was used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Duloxetine 60 mg
Number analyzed (Participants) | 149 | 146 | 153 | 149
percentage of participants | 22.8 | 28.8 | 23.5 | 37.6

6. Secondary Outcome: Change From Baseline in the Montgomery Åsberg Depression Rating Scale (MADRS) Total Score
Description: The MADRS is a depression rating scale consisting of 10 items, each rated 0 to 6. The 10 items represent the core symptoms of depressive illness. The overall score ranges from 0 (symptoms absent) to 60 (severe depression). A decrease in the total score or on individual items indicates improvement. LS means are from an ANCOVA model with treatment and center as fixed factors and the Baseline value as a covariate.
Time Frame: Baseline and Weeks 1, 2, 4, 6 and 8
Population: Full analysis set; LOCF was used. "n" indicates the number of patients included in the analysis at each time point.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Duloxetine 60 mg
Number analyzed (Participants) | 149 | 146 | 153 | 149
scores on a scale
  Week 1 (n=142, 143, 150, 147) | -4.90 (0.530) | -5.16 (0.511) | -5.06 (0.505) | -5.49 (0.514)
  Week 2 (n=149, 146, 153, 149) | -7.57 (0.615) | -7.71 (0.605) | -7.81 (0.599) | -8.95 (0.609)
  Week 4 (n=149, 146, 153, 149) | -9.66 (0.693) | -9.58 (0.681) | -9.35 (0.675) | -11.34 (0.686)
  Week 6 (n=149, 146, 153, 149) | -11.04 (0.770) | -11.25 (0.757) | -11.27 (0.750) | -13.29 (0.763)
  Week 8 (149, 146, 153, 149) | -11.22 (0.819) | -11.61 (0.805) | -11.30 (0.797) | -14.10 (0.811)

7. Secondary Outcome: Clinical Global Impression Scale-Global Improvement Scale
Description: The Clinical Global Impression - Global Improvement scale assesses the participant's improvement (or worsening) as assessed by the clinician relative to Baseline on a 7-point scale: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse. LS means were from an ANCOVA model with treatment and center as fixed factors and the CGI-S Baseline value as a covariate.
Time Frame: Baseline and Weeks 1, 2, 4, 6 and 8.
Population: Full analysis set; LOCF was used. "n" indicates the number of patients included in the analysis at each time point.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Duloxetine 60 mg
Number analyzed (Participants) | 149 | 146 | 153 | 149
scores on a scale
  Week 1 (n=142, 143, 149, 147) | 3.54 (0.067) | 3.42 (0.065) | 3.46 (0.064) | 3.31 (0.065)
  Week 2 (n=149, 146, 153, 149) | 3.21 (0.077) | 3.17 (0.076) | 3.10 (0.075) | 2.99 (0.076)
  Week 4 (149, 146, 153, 149) | 2.97 (0.085) | 2.93 (0.084) | 2.87 (0.083) | 2.73 (0.084)
  Week 6 (149, 146, 153, 149) | 2.83 (0.091) | 2.82 (0.090) | 2.74 (0.089) | 2.50 (0.090)
  Week 8 (n=149, 146, 153, 149) | 2.79 (0.098) | 2.73 (0.096) | 2.63 (0.095) | 2.39 (0.097)

8. Secondary Outcome: Change From Baseline in Montgomery-Åsberg Depression Rating Scale - Self-assessment (MADRS-S)
Description: The MADRS-S is a patient-reported outcome measure based on MADRS, administered to evaluate treatment effectiveness in depression. This scale consists of 9 items assessing patients' mood, feelings of unease, sleep, appetite, ability to concentrate, initiative, emotional involvement, pessimism and zest for life. Each item is scored between 0 (best) and 3 (worst). The total score is calculated by summing the answers of the nine items, ranging between 0 and 27 (higher scores indicate increased impairment). LS means are from an ANCOVA model with treatment and center as fixed factors and the Baseline value as a covariate.
Time Frame: Baseline and Weeks 1, 4 and 8
Population: Full analysis set with available data at Baseline; LOCF was used. "n" indicates the number of patients included in the analysis at each time point.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Duloxetine 60 mg
Number analyzed (Participants) | 148 | 145 | 152 | 149
scores on a scale
  Week 1 (n=141, 142, 149, 146) | -2.51 (0.310) | -2.43 (0.299) | -2.74 (0.295) | -2.88 (0.299)
  Week 4 (148, 145, 152, 149) | -4.02 (0.348) | -3.65 (0.342) | -3.69 (0.338) | -4.89 (0.342)
  Week 8 (n=148, 145, 152, 149) | -4.25 (0.370) | -3.98 (0.364) | -4.04 (0.360) | -5.70 (0.364)

9. Secondary Outcome: Change From Baseline in the Hamilton Anxiety Scale (HAM-A) Total Score
Description: The HAM-A is an anxiety rating scale consisting of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behavior at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total scores range from 0 to 56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe. Total scores above 30 are rare, but indicate very severe anxiety. LS means are from an ANCOVA model with treatment and center as fixed factors and the Baseline value as a covariate.
Time Frame: Baseline and Weeks 1, 2, 4, 6 and 8.
Population: Full analysis set; LOCF was used. "n" indicates the number of patients included in the analysis at each time point.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Duloxetine 60 mg
Number analyzed (Participants) | 149 | 146 | 153 | 149
scores on a scale
  Week 1 (n=142, 143, 150, 147) | -2.63 (0.356) | -2.98 (0.343) | -2.55 (0.339) | -2.30 (0.346)
  Week 2 (n=149, 146, 153, 149) | -3.82 (0.419) | -4.41 (0.412) | -3.76 (0.408) | -3.94 (0.415)
  Week 4 (n=149, 146, 153, 149) | -5.12 (0.457) | -5.10 (0.450) | -4.25 (0.445) | -4.88 (0.454)
  Week 6 (n=149, 146, 153, 149) | -5.84 (0.482) | -5.77 (0.474) | -4.89 (0.469) | -6.15 (0.478)
  Week 8 (n=149, 146, 153, 149) | -5.75 (0.502) | -5.91 (0.494) | -5.29 (0.488) | -6.56 (0.498)

10. Secondary Outcome: Change From Baseline in the Clinical Global Impression Scale-Severity of Illness Scale
Description: The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Considering total clinical experience, a patient is assessed on severity of mental illness on the following scale: 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill. LS means were from an ANCOVA model with treatment and center as fixed factors and the Baseline value as a covariate.
Time Frame: Baseline and Weeks 1, 2, 4, 6 and 8.
Population: Full analysis set; LOCF was used. "n" indicates the number of patients included in the analysis at each time point.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Duloxetine 60 mg
Number analyzed (Participants) | 149 | 146 | 153 | 149
scores on a scale
  Week 1 (n=142, 143, 150, 147) | -0.28 (0.055) | -0.40 (0.053) | -0.37 (0.053) | -0.44 (0.054)
  Week 2 (n=149, 146, 153, 149) | -0.63 (0.071) | -0.65 (0.069) | -0.66 (0.069) | -0.75 (0.070)
  Week 4 (n=149, 146, 153, 149) | -0.92 (0.086) | -0.92 (0.085) | -0.90 (0.084) | -1.12 (0.085)
  Week 6 (n=149, 146, 153, 149) | -1.11 (0.094) | -1.08 (0.092) | -1.08 (0.091) | -1.39 (0.093)
  Week 8 (n=149, 146, 153, 149) | -1.14 (0.103) | -1.21 (0.102) | -1.17 (0.101) | -1.56 (0.102)

11. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) Total Score at Week 8
Description: The Sheehan Disability Scale assesses functional impairment in 3 domains: work/school, social life or leisure activities, and home life or family responsibilities. The participant rates the extent to which each aspect is impaired on a 10-point visual analog scale, from 0 (not at all) to 10 (extremely). The 3 scores are added together to calculate the total score, which ranges from 0 to 30, with higher scores indicating more impairment. LS means were from an ANCOVA model with treatment and center as fixed factors and the Baseline value as a covariate.
Time Frame: Baseline and Week 8
Population: Full analysis set with available data at Baseline; LOCF was used.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Duloxetine 60 mg
Number analyzed (Participants) | 130 | 122 | 123 | 114
scores on a scale | -6.83 (0.638) | -6.46 (0.640) | -6.59 (0.641) | -8.91 (0.672)

12. Secondary Outcome: Healthcare Resource Utilization as Assessed by the Health Economic Assessment Questionnaire
Description: Healthcare resource utilization was assessed by the Health Economic Assessment (HEA) questionnaire, which monitors participants absenteeism from work, as well as resource use such as visits to a general practitioner, outpatient and inpatient services, hospitalization, medications, and other relevant services over the past 8 weeks.
Time Frame: Baseline and Week 8
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Duloxetine 60 mg
Number analyzed (Participants) | 149 | 146 | 153 | 149
participants
  Baseline: Any resource use | 40 | 51 | 42 | 42
  Baseline: Any hospitalization-related services | 4 | 1 | 0 | 3
  Baseline: Hospitalization related to depression | 2 | 1 | 0 | 0
  Baseline: Any sick leave | 18 | 11 | 11 | 14
  Baseline: Sick leave related to depression | 13 | 9 | 10 | 11
  Week 8: Any resource use | 21 | 19 | 20 | 27
  Week 8: Any hospitalization-related service | 1 | 0 | 1 | 2
  Week 8: Hospitalization related to depression | 0 | 0 | 0 | 1
  Week 8: Any sick leave | 5 | 5 | 9 | 5
  Week 8: Sick leave related to depression | 2 | 4 | 3 | 2

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the 8-week treatment period and a 4-week follow-up period.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Duloxetine 60 mg
Serious Adverse Events (participants affected / at risk) | 2/151 | 0/149 | 3/153 | 2/150
Other Adverse Events (participants affected / at risk) | 81/151 | 83/149 | 87/153 | 120/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=151) | Vortioxetine 2.5 mg (N=149) | Vortioxetine 5 mg (N=153) | Duloxetine 60 mg (N=150)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 1
Abortion induced (Surgical and medical procedures) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=151) | Vortioxetine 2.5 mg (N=149) | Vortioxetine 5 mg (N=153) | Duloxetine 60 mg (N=150)
Vision blurred (Eye disorders) | 3 | 1 | 1 | 4
Nausea (Gastrointestinal disorders) | 16 | 24 | 44 | 63
Dry mouth (Gastrointestinal disorders) | 11 | 16 | 16 | 40
Diarrhoea (Gastrointestinal disorders) | 13 | 7 | 14 | 19
Constipation (Gastrointestinal disorders) | 11 | 6 | 6 | 18
Vomiting (Gastrointestinal disorders) | 1 | 1 | 7 | 5
Dyspepsia (Gastrointestinal disorders) | 3 | 6 | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 6 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 0 | 5
Stomach discomfort (Gastrointestinal disorders) | 4 | 3 | 4 | 1
Flatulence (Gastrointestinal disorders) | 2 | 3 | 3 | 1
Fatigue (General disorders) | 5 | 3 | 3 | 13
Feeling jittery (General disorders) | 0 | 0 | 2 | 4
Irritability (General disorders) | 4 | 2 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 3 | 2 | 2 | 6
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 6 | 1 | 2
Weight decreased (Investigations) | 1 | 0 | 0 | 4
Blood pressure increased (Investigations) | 1 | 1 | 1 | 3
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 2 | 8
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 3 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 2 | 1 | 3
Headache (Nervous system disorders) | 18 | 20 | 24 | 21
Dizziness (Nervous system disorders) | 7 | 10 | 9 | 22
Somnolence (Nervous system disorders) | 6 | 3 | 9 | 20
Sedation (Nervous system disorders) | 4 | 3 | 5 | 1
Tension headache (Nervous system disorders) | 0 | 0 | 3 | 4
Tremor (Nervous system disorders) | 1 | 1 | 3 | 4
Insomnia (Psychiatric disorders) | 6 | 6 | 6 | 11
Restlessness (Psychiatric disorders) | 1 | 2 | 3 | 5
Anxiety (Psychiatric disorders) | 2 | 1 | 5 | 1
Libido decreased (Psychiatric disorders) | 3 | 3 | 3 | 4
Orgasm abnormal (Psychiatric disorders) | 0 | 0 | 3 | 3
Yawning (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 4 | 4 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.